CLINICAL TRIAL: NCT04852861
Title: COVID-19: Safety and Immunogenicity of a Reduced Dose of the BioNTech/Pfizer BNT162b2 Vaccine in a Healthy Population
Brief Title: COVID-19: Safety and Immunogenicity of a Reduced Dose of the BioNTech/Pfizer BNT162b2 Vaccine
Acronym: REDU-VAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sciensano (Other Government)
Collaborators: Mensura EDPB (Unknown); Institute of Tropical Medicine, Belgium (Other); Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Maria Goossens, Scientific collaborator, Sciensano
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DemiVac2021; 2021-002088-23 (EudraCT Number)
Record Dates: First submitted 2021-04-14; First posted 2021-04-21 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: vaccination; Covid19; immunogenicity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research nurse administrating the vaccine is the only one who is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comirnaty®; Pfizer-BioNTech BNT162b2 mRNA 20 mcg (Experimental): In this arm participants will receive two doses of Comirnaty BNT162b2 mRNA 20 mcg.
  Interventions: Diagnostic Test: immunogenicity after first and second dose
- Comirnaty®; Pfizer-BioNTech BNT162b2 mRNA 30 mcg (Active Comparator): In this arm participants will receive two doses of Comirnaty BNT162b2 mRNA 30 mcg.
  Interventions: Diagnostic Test: immunogenicity after first and second dose

INTERVENTIONS:
Diagnostic Test: immunogenicity after first and second dose — Humoral and cellulair immunity after first and second dose of the different vaccines administrated.

SUMMARY:
This is a randomized phase IV dose-optimization study evaluating the safety and immunogenicity of two doses of COVID-19 mRNA vaccines being authorized in the European Union since December 2020: Vaccine BNT162b2 (Comirnaty®; Pfizer-BioNTech) in healthy adults up to age 55 year. Immunogenicity will be measured 28 days after first and second dose, and day 180 and day 365 after first vaccination of 20 and 30 mcg of BNT162b2. The primary outcome is the level of binding antibodies for RBD 28 days after the second dose.

DETAILED DESCRIPTION:
Background: Data from the dose-escalating phase 1 trials from the COVID-19 mRNA vaccines being authorized in the European Union since December 2020, BNT162b2 (Comirnaty®; Pfizer- BioNTech) indicate that for the age group 18-55 years a lower dose of the vaccine can induce the same immune response as the full dose.

Method: This is a randomized multicenter phase IV dose-optimization study evaluating the safety and immunogenicity of demi-doses of a COVID-19 mRNA vaccine being authorized in the European Union since December 2020, BNT162b2 (Comirnaty®; Pfizer- BioNTech) in healthy adults up to age 55 year. The study will be performed in employees of Mensura EDPB at five different sites.

Objectives: The primary outcome is the level of binding antibodies for RBD 28 days after the second dose. Secondary outcomes are safety and reactogenicity after vaccination. The neutralizing antibodies and the cellular immunity 28 days after second dose will be assessed. Humoral and cellular immunity will be measured 180 and 365 days after first dose.

ELIGIBILITY:
Inclusion Criteria: Working at Mensura EDPB, not yet vaccinated for COVID19 -

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titre (GMT) of Binding antibodies to the RBD of SARS-CoV-2 S protein | 28 days after second dose
  Binding antibodies anti-RBD

SECONDARY OUTCOMES:
GMT of Neutralizing anti-bodies to Wuhan strain and variants | 28 days after second dose
T cell response to S protein of Wuhan strain and variants and Memory B cell responses to S protein of Wuhan strain and variants | 28 days after second dose
Humoral and cellulair immunity | 180 days after first dose
  GMT of of Binding antibodies to the RBD of SARS-CoV-2 S protein and Neutralizing anti-bodies to Wuhan strain and variants and T cell response to S protein of Wuhan strain and variants and Memory B cell responses to S protein of Wuhan strain and variants
Humoral and cellulair immunity | 365 days after first dose
  GMT of of Binding antibodies to the RBD of SARS-CoV-2 S protein and Neutralizing anti-bodies to Wuhan strain and variants and T cell response to S protein of Wuhan strain and variants and Memory B cell responses to S protein of Wuhan strain and variants
safety and reactogenicity | through study completion, an average of 1 year
  adverse events will be followed up after vaccine adminstration

CONTACTS AND LOCATIONS:
Locations (1):
- Mensura EDPB, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pannus P, Depickere S, Kemlin D, Houben S, Neven KY, Heyndrickx L, Michiels J, Willems E, De Craeye S, Francotte A, Chaumont F, Olislagers V, Waegemans A, Verbrugghe M, Schmickler MN, Van Gucht S, Dierick K, Marchant A, Desombere I, Arien KK, Goossens ME. Safety and immunogenicity of a reduced dose of the BNT162b2 mRNA COVID-19 vaccine (REDU-VAC): A single blind, randomized, non-inferiority trial. PLOS Glob Public Health. 2022 Dec 20;2(12):e0001308. doi: 10.1371/journal.pgph.0001308. eCollection 2022. PMID 36962838